CLINICAL TRIAL: NCT00947362
Title: Phase 2 Study Electrothermocauterisation of Afghan Patients With Anthroponotic Cutaneous Leishmaniasis With and Without Pharmaceutical Chlorite Listed in the German Drug Codex (DAC N-055)
Brief Title: Rationale for New Topical Anthroponotic Cutaneous Leishmaniasis (ACL) Treatment in Kabul
Acronym: rtt-ACL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Waisenmedizin e. V. Promoting Access to Essential Medicine (Other)
Collaborators: German Medical Service (GMS) in Kabul (Other); University of Freiburg (Other)
Responsible Party: Principal Investigator, Kurt-Wilhelm Stahl, Chairman, Waisenmedizin e. V. Promoting Access to Essential Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 169/04; No grant or contract number
Record Dates: First submitted 2009-07-24; First posted 2009-07-28 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Wound Healing
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ETC + DAC N-055 (Experimental)
  Interventions: Other: Electro-thermo-coagulation; Drug: DAC N-055
- ETC + physiological saline (Active Comparator)
  Interventions: Other: Electro-thermo-coagulation; Drug: saline

INTERVENTIONS:
Other: Electro-thermo-coagulation
Drug: DAC N-055 — moist wound treatment plus 0.05 % pharmaceutical chlorite
  Arms: ETC + DAC N-055
Drug: saline — physiological saline
  Arms: ETC + physiological saline

SUMMARY:
The aim of the randomized double blind trial with 134 patients presenting old world cutaneous leishmaniasis is:

* to evaluate the clinical efficacy of electro-thermo-cauterisation (ETC) followed by moist wound treatment versus ETC followed by moist wound treatment plus 0.05 % pharmaceutical chlorite that has been used in three European countries (Germany, Austria and Switzerland) in wound care management for more than 20 years;
* to judge whether early wound care management would present a viable improvement to the actual anti-parasitic treatments mostly neglecting the chronic wound problem and to evaluate its long-term effect on immunity through relapse control 6 months after wound healing.

ELIGIBILITY:
Inclusion Criteria:

* at least one suspected lesion positive in Giemsa smear

Exclusion Criteria:

* patients previously treated for leishmania

Ages: 5 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2004-08-01 (Actual); Primary Completion 2007-12-15 (Actual); Study Completion 2007-12-15 (Actual)

PRIMARY OUTCOMES:
Days for wound closure | From the day of treatment start to the day of "wound closure"
  Days for primary wound closure

SECONDARY OUTCOMES:
Leishmania parasites load per gram of tissue before and after treatment | Before treatment start and at day "wound closure"
  Parasite load per gram of tissue

CONTACTS AND LOCATIONS:
Locations (1):
- German Medical Service, Kabul, Kabul, Afghanistan

REFERENCES:
- [Derived] Jebran AF, Schleicher U, Steiner R, Wentker P, Mahfuz F, Stahl HC, Amin FM, Bogdan C, Stahl KW. Rapid healing of cutaneous leishmaniasis by high-frequency electrocauterization and hydrogel wound care with or without DAC N-055: a randomized controlled phase IIa trial in Kabul. PLoS Negl Trop Dis. 2014 Feb 13;8(2):e2694. doi: 10.1371/journal.pntd.0002694. eCollection 2014 Feb. PMID 24551257